CLINICAL TRIAL: NCT07236099
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study of the Efficacy and Safety of ICP-332 in Participants With Prurigo Nodularis
Brief Title: Study of the Efficacy and Safety of ICP-332 in Participants With Prurigo Nodularis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICP-CL-00609
Record Dates: First submitted 2025-10-27; First posted 2025-11-19 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Prurigo Nodularis (PN)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ICP-332 80mg (Experimental)
  Interventions: Drug: ICP-322
- ICP-332 120mg (Experimental)
  Interventions: Drug: ICP-322
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ICP-322 — ICP-322 Tablets
  Arms: ICP-332 120mg; ICP-332 80mg
Drug: Placebo — ICP-332 Placebo Tablets
  Arms: Placebo

SUMMARY:
Evaluate the efficacy and safety of ICP-332 in participants with Prurigo Nodularis (PN)

ELIGIBILITY:
Inclusion Criteria :

1. Voluntarily sign informed consent forms before any investigational procedure(s) are performed.
2. Male or female aged between 18 and 75 years at the time of signing the informed consent.
3. Clinical diagnosis of PN by a dermatologist for at least 3 months before the Screening visit.
4. At least 20 pruriginous lesions on the entire body with a bilateral distribution (on both legs, and/or both arms and/or trunk) at both screening and the baseline (Day 1) visits.
5. PP NRS score ≥ 7 at both screening and the baseline (Day 1) visits.
6. IGA-CPG-S score ≥ 3 at both the screening and the baseline (Day 1) visits.
7. History of inadequate response to topical corticosteroid of medium or higher potency or for whom topical treatments are otherwise medically inadvisable (e.g., because of important side effects or safety risks).

Willingness to avoid pregnancy or fathering children

Exclusion Criteria:

1. Patients with a documented AD severity moderate to severe presence of skin morbidities other than PN and mild AD that may interfere with the assessment of the study outcomes. PN secondary to medications .
2. Any uncontrolled or serious disease, or any medical, psychological, or surgical condition including relevant laboratory abnormalities at screening that may either interfere with the interpretation of the clinical trial results and/or, in the investigator's judgment, would adversely affect the patient's participation in the study. Active chronic or acute infection participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Peak pruritus-numeric rate scale (PP NRS) | Baseline to week 16
  Percent change from baseline of weekly average in Peak pruritus-numeric rate scale (PP NRS) at Week 16. Participants will be asked to rate their itch at the worst moment during the previous 24 hours. On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable'.

SECONDARY OUTCOMES:
Improvement in PP NRS score | Baseline through week 40
  Proportion of participants achieving ≥ 4-point improvement in PP NRS score (PP NRS ≥ 4) over time
Investigator's Global Assessment for Chronic Prurigo Stage scores of 0 or 1 (IGA-CPG-S 0/1) | Baseline through week 40
  Proportion of participants achieving Investigator's Global Assessment for Chronic Prurigo Stage scores of 0 or 1 (IGA-CPG-S 0/1) over time
Dermatology Life Quality Index (DLQI) | Baseline through week 40
  Change from baseline in Dermatology Life Quality Index (DLQI) score over time. The DLQI comprises 10 items assessing the impact of skin disease on patients' health-related quality of life (HRQoL) over the previous week. Overall scoring ranges from 0 to 30, with a high score indicative of a poor HRQoL
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Baseline through week 40
Maximum concentration (Cmax) | Baseline through week 40
  Maximum concentration (Cmax) of ICP-322
Area Under Concentration Versus Time Curve (AUC) | Baseline through week 40
  Area Under Concentration Versus Time Curve (AUC) of ICP-322

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - The Second Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The first hospital of Jilin University, Changchun, Jilin
  - Shenyang Seventh People's Hospital, Shenyang, Liaoning
  - Shandong Provincial Dermatology Hospital, Jinan, Shandong
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - Affiliated Hangzhou First People's Hospital,School of Medicine ,Westlake University, Hangzhou, Zhejiang